CLINICAL TRIAL: NCT06818123
Title: Exploring the Effectiveness of Interventions on Menstrual Hygiene Awareness in Slum Communities of Karachi, A Quasi- Experimental Analysis.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SINA Health Education and Welfare Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0006
Record Dates: First submitted 2024-09-28; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Menstruations; Menstruation Hygiene; Hygiene Practices and Knowledge; Knowledge Gaps; Social Stigma
Keywords: Hygiene Practice; Slums Area; Knowledge and practices; Knowledge Gaps; Poor Hygiene; Menstruation Hygiene
MeSH Terms: conditions — Social Stigma | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (Placebo Comparator): Education Intervention along with the doctor's consultation
  Interventions: Other: Control group with doctor's consultation only
- Intervention (Experimental): Those who will be under the baseline screening in term of knowledge, will then treated as interventional arm and interventional will be given to them.
  Interventions: Other: Education Intervention along with the doctor's consultation

INTERVENTIONS:
Other: Education Intervention along with the doctor's consultation — This educational intervention will assess the improvement menstrual hygiene knowledge and practices among women at slums who are illiterate and can empower individuals to manage their periods with dignity and comfort.
  Arms: Intervention
Other: Control group with doctor's consultation only — Baseline Knowledge will be assessed in this arm about the menstruations hygiene and practices.
  Arms: Control Arm

SUMMARY:
Proper menstrual hygiene knowledge and practices are crucial among women. People of urban slum's areas have no or less knowledge and practices of Menstruation hygiene due to low socio-economic status. This study helps in Improving menstrual hygiene knowledge and practices and can empower individuals to manage their periods with dignity and comfort. This study also contributes in creating a more open and supportive environment for menstruation by addressing stigma and misconception. The study also helps in reducing the risk of reproductive tract infections.

ELIGIBILITY:
Inclusion Criteria:

* Woman age in between 15-45years of age
* Those who used reusable items for menstruations
* Those who are willing to participate voluntarily will be included in the study

Exclusion Criteria:

* Participants who are suffering from any serious medical condition.
* live in other than slums area of Karachi will be excluded from the study.

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — The study is to check menstruations hygiene knowledge among women at slums. Menstruations hygiene knowledge can only be check in women without menopause and who are in age of puberty
Enrollment: 400 (Estimated)
Dates: Start 2025-02-28 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Improved Menstruations Hygiene knowledge | one month
  Effectiveness of educational intervention of menstruation hygiene among participants

SECONDARY OUTCOMES:
Reduction in vaginal infection | one month
  Recurrent Infection such as yeast infection, discomfort, itching, other related infection.
promoting better self-esteem and confidence | one month
  Participants who is taking the education session and counselling, adapt the good women hygiene

CONTACTS AND LOCATIONS:
Locations (1):
- SINA Health Education and Welfare Trust, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No